CLINICAL TRIAL: NCT04005612
Title: Assessing the Combined Effect of Omega-3 Fatty Acid and Vitamin D3 on Plasma Osteocalcin Levels : a Randomized Controlled Trial in Males and Females With Vitamin D Deficiency
Brief Title: Effect of Vitamin d and Omega 3 on Osteocalcin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science Private University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DRGS-2014-2015-165-3
Record Dates: First submitted 2019-07-01; First posted 2019-07-02 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D Deficiency; plama osteocalcin; omega-3 fatty acids
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Fatty Acids, Omega-3

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- vitamin d3 group (Experimental): weekly Dietary Supplement: Vitamin D3 50,000 IU Vitamin D3 / week for 8 weeks
  Interventions: Dietary Supplement: vitamin D3; Dietary Supplement: omega-3 fatty acid; Dietary Supplement: vitamin D3 and omega-3 fatty acid; Other: control
- omega3-Fatty Acid group (Experimental): 1000 mg wild salmon and fish oil complex (contains 300 mg of omega3-FA) once daily
  Interventions: Dietary Supplement: vitamin D3; Dietary Supplement: omega-3 fatty acid; Dietary Supplement: vitamin D3 and omega-3 fatty acid; Other: control
- VD3 and Omega-3FA group (Experimental): 50,000 IU VD3 / week and 1000 mg wild salmon and fish oil complex (contains 300 mg of omega-3 FA) once daily
  Interventions: Dietary Supplement: vitamin D3; Dietary Supplement: omega-3 fatty acid; Dietary Supplement: vitamin D3 and omega-3 fatty acid; Other: control
- Control group (No Intervention): NO INTERVENTION

INTERVENTIONS:
Dietary Supplement: vitamin D3 — 50,000 IU VD3 / week for 8 weeks
  Arms: VD3 and Omega-3FA group; omega3-Fatty Acid group; vitamin d3 group
Dietary Supplement: omega-3 fatty acid — 300 mg of omega 3-FA once daily for 8 weeks
  Arms: VD3 and Omega-3FA group; omega3-Fatty Acid group; vitamin d3 group
Dietary Supplement: vitamin D3 and omega-3 fatty acid — 50,000 IU VD3 / week for 8 weeks and 300 mg of omega-3FA once daily for 8 weeks
  Arms: VD3 and Omega-3FA group; omega3-Fatty Acid group; vitamin d3 group
Other: control — no intervention
  Arms: VD3 and Omega-3FA group; omega3-Fatty Acid group; vitamin d3 group

SUMMARY:
Assessing the combined effect of omega-3 fatty acid and vitamin D 3 on plasma osteocalcin levels

DETAILED DESCRIPTION:
The data about effect of vitamin D3 (VD3) and omega-3 fatty acids(omega-3FA) on plasma levels of osteocalcin (OCN) are scarce and conflicting and nothing is published in the literature about the effect of the combination of VD3 and omega-3FA on the OCN levels.

This study was conducted to investigate effect of VD3 and omega-3FA alone and with each other on PLASMA OCN levels in females and males with vitamin D deficiency (VDD).

This randomized, controlled clinical trial was designed to test effects of 50,000 IU VD3 weekly and 300 mg omega-3FA daily for eight weeks,separately and with each other, on the plasma levels of OCN and 25-hydroxy vitamin D (25OHD).

This study was conducted during winter in 86 healthy Jordanian females and males with VDD with a mean age of (40± 10) years.

Fasting serum levels for 25OHD,OCN, PTH (parathyroid hormone),calcium, phosphate, ALT (alanine aminotransferase), and urea were assessed at baseline and the end of the trial .

ELIGIBILITY:
Inclusion Criteria:

* Medical diagnosis of vitamin D deficiency (VD < 30 ng / ml).

Exclusion Criteria:

* People who previously diagnosed with any chronic disease such as kidney diseases were excluded from the study due to the effect of prolonged administration of VD3 on kidney stones formation.
* People with bone disorders also excluded.

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
vitamin d3 levels | 8 weeks
  Plasma levels of 25-hydroxyvitamin D
osteocalcin levels | 8 weeks
  plasma osteocalcin levels

SECONDARY OUTCOMES:
PTH | 8 weeks
  Plasma concentrations of PTH
calcium | 8 weeks
  plasma Ca levels

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S Abu-Samak, PhD, Principal Investigator — Applied Science Private University
Locations (1):
- Applied Science University, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: when summary data are published
Access Criteria: open access

REFERENCES:
- [Background] Holick MF, Chen TC. Vitamin D deficiency: a worldwide problem with health consequences. Am J Clin Nutr. 2008 Apr;87(4):1080S-6S. doi: 10.1093/ajcn/87.4.1080S. PMID 18400738